CLINICAL TRIAL: NCT01652573
Title: Calcitonin for Treating X-linked Hypophosphatemia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Yale University (Other)
Collaborators: National Institute of Arthritis and Musculoskeletal and Skin Diseases (NIAMS) (NIH)
Responsible Party: Principal Investigator, Karl Insogna, Professor of Medicine, Yale University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 1010007548; R21AR061818 (NIH)
Record Dates: First submitted 2012-07-23; First posted 2012-07-30 (Estimated); Results first posted 2017-05-31 (Actual); Last update posted 2017-05-31 (Actual); Status verified 2017-04

CONDITIONS: Hypophosphatemic Rickets, X Linked Dominant
Keywords: X linked hypophosphatemia; calcitonin; FGF twenty three
MeSH Terms: conditions — Familial Hypophosphatemic Rickets | interventions — salmon calcitonin

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Nasal calictonin (Experimental): Subjects will received nasal calcitonin once daily
  Interventions: Drug: nasal salmon calcitonin
- Saline Nasal spray (Placebo Comparator): Patients will receive saline nasal spray once daily
  Interventions: Drug: Saline Nasal Spray Placebo

INTERVENTIONS:
Drug: nasal salmon calcitonin — 400 IU daily in two sprays (one to each nares)
  Other Names: Miacalcin; Fortical
  Arms: Nasal calictonin
Drug: Saline Nasal Spray Placebo
  Arms: Saline Nasal spray

SUMMARY:
X-linked hypophosphatemia (XLH) is the most common form of inherited rickets in the United States. It also causes bone disease in adults. XLH is caused by overproduction of a hormone call FGF23, which makes the body waste phosphate. This study is designed to determine if nasal calcitonin, an already approved drug in the US, can lower blood levels of FGF23 and reduce phosphate wasting in patients with XLH. In this study the investigators will:

1. Determine whether nasal calcitonin significantly lowers integrated 24-hour blood levels of FGF23 in patients with XLH.
2. Evaluate whether nasal calcitonin improves serum phosphate levels in XLH.
3. Assess whether nasal calcitonin improves blood levels of the active form of vitamin D and calcium absorption from the intestine.
4. Make sure that nasal calcitonin is safe and well tolerated.

DETAILED DESCRIPTION:
The pathophysiology of X-linked hypophosphatemia (XLH) was clarified with the report in 1995 by the HYP Consortium led by Dr. Michael Econs, that mutations in the neutral endopeptidase PHEX, are the genetic basis for this disorder (Nature Genetics 11:130). By a pathway that remains unclear, loss-of-function mutations in PHEX lead to elevated circulating levels of FGF23. It is now well established that FGF23 is the proximate biological mediator of this syndrome. FGF23 suppresses renal tubular phosphate reabsorption by inhibiting transcription of the major sodium phosphate co-transporters in the proximal renal tubule. In addition, it suppresses 1-α hydroxylase activity leading low to low-normal serum levels of 1,25(OH)2vitamin D. This in turn impairs intestinal phosphate and calcium absorption. These combined biochemical abnormalities lead to persistent defects in skeletal mineralization manifested as rickets in children and osteomalacia in adults. Conventional therapy for XLH consists of oral therapy with phosphate supplements and calcitriol and requires ingestion of medications 4-6 times daily. There are several limitations to conventional therapy including its inability to correct growth retardation in children or the enthesopathy so frequently seen in adults. Furthermore, it is now clear that this therapeutic approach causes a further rise in circulating levels of FGF23 in XLH. Thus, there is an urgent need for more appropriate therapy directed at the basic pathophysiology of this disorder. As detailed in the Research Strategy, we have identified calcitonin as a novel suppressor of FGF23 production in XLH. A single, subcutaneous injection of calcitonin results in a sustained fall in FGF23 levels that persists for 16 hours after drug administration; a change not observed in control subjects. The fall in serum FGF23 is associated with a rise in serum phosphate and circulating levels of 1,25(OH)2vitamin D. These data are very exciting as they suggest a novel therapy for XLH. This exploratory clinical trial seeks to establish the efficacy of calcitonin in improving the biochemical abnormalities in untreated adults with XLH. We will test the hypothesis that calcitonin, by lowering circulating levels of FGF23 and raising serum levels of 1,25(OH)2vitamin D, will improve phosphate homeostasis in patients with XLH. To test this hypothesis we will pursue the following specific aims: 1. Determine whether 3 months of nasal calcitonin administered at a dose of 400 IU/day significantly lowers integrated 24-hour serum levels of FGF23 in patients with XLH. 2. Evaluate whether nasal calcitonin improves phosphate homeostasis by raising the TmP/GFR and integrated 24 hr. serum phosphate concentrations. 3. Assess whether nasal calcitonin improves calcium metabolism in patients with XLH by increasing integrated 24 hr. serum levels of 1,25(OH)2vitamin D and enhancing intestinal calcium absorption, as estimated by 24-hour urine calcium. 4. Confirm that nasal calcitonin is well tolerated by quantifying side effects and nasal irritation during the trial.

If successful, this study will provide proof-of-principal for the novel use of an FDA-approved drug in treating XLH. This approach, unlike conventional treatment, addresses the underlying pathophysiology in this disorder and would represent the first therapeutic advance for XLH in 30 years.

ELIGIBILITY:
Inclusion Criteria:

* age ≥18 or greater
* an established diagnosis of XLH
* fasting serum calcium ≤10.5 mg/dl
* fasting PTH at time of screen </= 1.7 times the upper limit of normal

Exclusion Criteria:

* estimated creatinine clearance < 60 cc/min and/or serum creatinine > 1.5 mg/dl;
* serum 25(OH)vitamin D < 30 ng/ml. Potential study subjects who have a serum 25(OH)vitamin D < 30 ng/ml will be supplemented with 25(OH)vitamin D to achieve a serum value > 30 ng/ml and then re- screened
* inability to comply with instructions and appropriate follow up visits
* treatment with agents that may skeletal metabolism such as glucocorticoids, bisphosphonates, denosumab, teriparatide, estrogen and anticonvulsants.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2011-03; Primary Completion 2015-09 (Actual); Study Completion 2015-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Karl L Insogna, MD, Principal Investigator — Profossor of Medicine, Yale School of Medicine
Locations (1):
- Yale School of Medicine, New Haven, Connecticut, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects were recruited from the individual practices of two of the physicians on this study and from a panel of patients with XLH who had previously participated or inquired about participation in ongoing clinical trials at this institution.
Pre-assignment Details: Patients who were receiving conventional therapy with calcitriol and phosphorus at the time of screening were asked to stop both agents two weeks prior to enrolling in the study and no subjects took calcitriol or phosphorus during the entire study.
Groups:
- Saline Nasal Spray: Patients will receive saline nasal spray once daily
  Saline Nasal Spray Placebo
Period: Overall Study
Arm/Group | Nasal Calictonin | Saline Nasal Spray
Started | 10 | 11
Completed | 10 | 10
Not Completed | 0 | 1
Not completed — Adverse Event | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Nasal Calictonin | Saline Nasal Spray | Total
Number analyzed (Participants) | 10 | 11 | 21
Age, Continuous [Mean (Full Range); unit: years] | 47 [26 to 66] | 47 [32 to 64] | 47 [26 to 66]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9 | 7 | 16
  Male | 1 | 4 | 5
Region of Enrollment [Number; unit: participants]
  United States | 10 | 11 | 21

OUTCOME MEASURES:

1. Primary Outcome: Area Under the Curve for FGF23
Description: FGF23 will be measured 0 to 24 hours post dose during a 24 hour admission and AUC calculated.
Time Frame: Time 0
Measure: Least Squares Mean (95% Confidence Interval); unit: pg/ml*hr
Arm/Group | Nasal Calictonin | Saline Nasal Spray
Number analyzed (Participants) | 10 | 11
pg/ml*hr | 3172.34 [3068.7 to 3332.68] | 3215.34 [3107.17 to 3374.97]

2. Primary Outcome: Area Under the Curve for FGF23
Description: FGF23 will be measured 0 to 24 hours post dose during a 24 hour admission at 3 months and AUC calculated and compared to baseline.
Time Frame: 3 months
Measure: Least Squares Mean (95% Confidence Interval); unit: pg/ml*hr
Arm/Group | Nasal Calictonin | Saline Nasal Spray
Number analyzed (Participants) | 10 | 11
pg/ml*hr | 2698.38 [2623.07 to 2830.39] | 2994.26 [2907.61 to 3134.26]

3. Secondary Outcome: Area Under the Curve for TmP/GFR
Description: Serum phosphate will be measured 0 to 24 hours postdose during a 24 hr admission, AUC calculated, and fasting Tmp/GFR calculated.
Time Frame: Time 0
Measure: Least Squares Mean (95% Confidence Interval); unit: mg/100 ml GF*hr
Arm/Group | Nasal Calictonin | Saline Nasal Spray
Number analyzed (Participants) | 10 | 11
mg/100 ml GF*hr | 30.70 [29.5 to 32.27] | 29.97 [28.78 to 31.49]

4. Secondary Outcome: Area Under the Curve for 1,25(OH)2vitamin D
Description: Serum 1,25(OH)2vitamin D will be measured 0 to 24 hours post dose during a 24 hr admission and AUC calculated.
Time Frame: Time 0
Measure: Least Squares Mean (95% Confidence Interval); unit: ng/ml*hr
Arm/Group | Nasal Calictonin | Saline Nasal Spray
Number analyzed (Participants) | 10 | 11
ng/ml*hr | 904.06 [862.86 to 961.90] | 838.58 [799.18 to 892.99]

5. Secondary Outcome: Number of Patients With Nasal Congestion at Baseline
Description: This symptom will be assessed at baseline
Time Frame: Time 0
Measure: Count of Participants; unit: Participants
Arm/Group | Nasal Calictonin | Saline Nasal Spray
Number analyzed (Participants) | 10 | 11
Participants | 0 | 0

6. Secondary Outcome: Area Under the Curve for TmP/GFR
Description: TmP/GFR will be measured 0 to 24 hours postdose during a 24 hr admission at 3 months and AUC calculated and compared to baseline.
Time Frame: Time 3 months
Measure: Least Squares Mean (95% Confidence Interval); unit: mg/100 ml GF*hr
Arm/Group | Nasal Calictonin | Saline Nasal Spray
Number analyzed (Participants) | 10 | 11
mg/100 ml GF*hr | 32.17 [31.04 to 33.68] | 31.26 [30.13 to 32.74]

7. Secondary Outcome: Area Under the Curve for 1,25(OH)2vitamin D
Description: Serum 1,25(OH)2vitamin D will be measured 0 to 24 hours post dose during a 24 hr admission and AUC calculated and results will be compared to baseline values.
Time Frame: Time 3 months
Measure: Least Squares Mean (95% Confidence Interval); unit: ng/ml*hr
Arm/Group | Nasal Calictonin | Saline Nasal Spray
Number analyzed (Participants) | 10 | 11
ng/ml*hr | 1277.05 [1235.72 to 1335.02] | 1258.84 [1217.74 to 1315.70]

8. Secondary Outcome: Number of Participants With Nasal Congestion at 1 Month
Description: This symptom will be assessed.
Time Frame: Time 1 month
Measure: Count of Participants; unit: Participants
Arm/Group | Nasal Calictonin | Saline Nasal Spray
Number analyzed (Participants) | 10 | 11
Participants | 3 | 2

9. Secondary Outcome: Number of Participants With Nasal Congestion at 2 Months
Description: This symptom will be assessed.
Time Frame: Time 2 months
Measure: Count of Participants; unit: Participants
Arm/Group | Nasal Calictonin | Saline Nasal Spray
Number analyzed (Participants) | 10 | 10
Participants | 1 | 0

10. Secondary Outcome: Number of Participants With Nasal Congestion at 3 Months
Description: This symptom will be assessed.
Time Frame: Time 3 months
Measure: Count of Participants; unit: Participants
Arm/Group | Nasal Calictonin | Saline Nasal Spray
Number analyzed (Participants) | 10 | 10
Participants | 0 | 0

11. Secondary Outcome: Number of Participants With Nasal Ulcerations at Baseline
Description: This symptom will be assessed at baseline
Time Frame: Time 0
Measure: Count of Participants; unit: Participants
Arm/Group | Nasal Calictonin | Saline Nasal Spray
Number analyzed (Participants) | 10 | 11
Participants | 0 | 0

12. Secondary Outcome: Number of Participants With Allergic Reactions at Baseline
Description: This symptom will be assessed at baseline
Time Frame: Time 0
Measure: Count of Participants; unit: Participants
Arm/Group | Nasal Calictonin | Saline Nasal Spray
Number analyzed (Participants) | 10 | 11
Participants | 0 | 0

13. Secondary Outcome: Number of Participants With Nasal Ulceration at 1 Month
Description: This symptom will be assessed.
Time Frame: Time 1 month
Measure: Count of Participants; unit: Participants
Arm/Group | Nasal Calictonin | Saline Nasal Spray
Number analyzed (Participants) | 10 | 11
Participants | 0 | 2

14. Secondary Outcome: Number of Participants With Allergic Reactions at 1 Month
Description: This symptom will be assessed.
Time Frame: Time 1 month
Measure: Count of Participants; unit: Participants
Arm/Group | Nasal Calictonin | Saline Nasal Spray
Number analyzed (Participants) | 10 | 11
Participants | 0 | 0

15. Secondary Outcome: Number of Participants With Nasal Ulceration at 2 Months
Description: This symptom will be assessed.
Time Frame: Time 2 months
Measure: Count of Participants; unit: Participants
Arm/Group | Nasal Calictonin | Saline Nasal Spray
Number analyzed (Participants) | 10 | 10
Participants | 0 | 0

16. Secondary Outcome: Number of Participants With Allergic Reactions at 2 Months
Description: This symptom will be assessed.
Time Frame: Time 2 months
Measure: Count of Participants; unit: Participants
Arm/Group | Nasal Calictonin | Saline Nasal Spray
Number analyzed (Participants) | 10 | 10
Participants | 0 | 0

17. Secondary Outcome: Number of Participants With Nasal Ulcerations at 3 Months
Description: This symptom will be assessed.
Time Frame: Time 3 months
Measure: Count of Participants; unit: Participants
Arm/Group | Nasal Calictonin | Saline Nasal Spray
Number analyzed (Participants) | 10 | 10
Participants | 0 | 1

18. Secondary Outcome: Number of Participants With Allergic Reactions at 3 Months
Description: This symptom will be assessed.
Time Frame: Time 3 months
Measure: Count of Participants; unit: Participants
Arm/Group | Nasal Calictonin | Saline Nasal Spray
Number analyzed (Participants) | 10 | 10
Participants | 0 | 0

ADVERSE EVENTS:
Time Frame: Adverse events were collected from the baseline visit until the end of study at 3 months.
Arm/Group | Nasal Calictonin | Saline Nasal Spray
All-Cause Mortality (participants affected / at risk) | 0/10 | 0/11
Serious Adverse Events (participants affected / at risk) | 0/10 | 0/11
Other Adverse Events (participants affected / at risk) | 2/10 | 2/11
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Nasal Calictonin (N=10) | Saline Nasal Spray (N=11)
Dermatologic (Skin and subcutaneous tissue disorders) | 1 (1) | 2 (2)
musculoskeletal events (Musculoskeletal and connective tissue disorders) | 1 (1) | 2 (2)
Respiratory events (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 2 (2)

LIMITATIONS AND CAVEATS:
It is possible that there is a threshold serum concentration of drug required to suppress FGF23 levels and our sample size was small.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No